CLINICAL TRIAL: NCT06396273
Title: Vision-Based Assessment of Driving Ability in Individuals With Dementia
Brief Title: Eye Scanning for Safety Driving
Status: Active, not recruiting | Type: Observational
Sponsor: Loughborough University (Other)
Collaborators: Monash University (Other)
Responsible Party: Principal Investigator, Ahmet Begde, Research Associate, Loughborough University
Other Study IDs: LoughboroughUn
Record Dates: First submitted 2024-04-25; First posted 2024-05-02 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Dementia; Mild Cognitive Impairment; Older Adults
MeSH Terms: conditions — Dementia; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- participants with cognitive impairment aged 65
- older adults without cognitive impairment

SUMMARY:
This is an experimental study protocol to investigate the use of vision-based assessments like eye-tracking and visual processing tests to evaluate driving ability in older adults with and without dementia. The study aims to address the research gap on the specific eye movement patterns and visual behaviors of individuals with Alzheimer's disease during high-risk driving scenarios.

The study will recruit 15 participants aged 65+ with cognitive impairment and 15 without cognitive impairment. Their cognitive status will be assessed using the Mini-Mental State Exam (MMSE) and Hopkins Verbal Learning Test (HVLT). Participants will undergo visual screening tests like visual sensitivity, eye movement scanning, and the Corsi block span test. Their driving performance will be evaluated through a hazard perception test and driving experience survey.

Statistical analyses like correlations, group comparisons, regression, and mediation analyses will be conducted to examine the relationships between cognitive status, visual screening scores, and driving performance scores. The goal is to determine if visual measures can predict driving ability and mediate the link between cognitive function and driving performance in those with dementia.

In summary, it is a protocol for an observational study using vision-based techniques to assess driving capacity in older adults, especially those with Alzheimer's disease or dementia.

ELIGIBILITY:
Inclusion Criteria:

* Participants with cognitive impairment aged 65 and/or older and older adults without cognitive impairment will be recruited for this study.

Exclusion Criteria:

* Participants with other neurological disease (stroke, Parkinson's, or multiple sclerosis),
* Psychiatric conditions (depression, anxiety disorder, etc.) and a history of severe psychiatric disorders (schizoaffective/bipolar disorders, or schizophrenia),
* Severe vision/hearing impairments that cannot be corrected with aids,
* Unable to comprehend questionnaire material study procedures and give consent.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: participants with cognitive impairment aged 65 and/or older and 20 older adults without cognitive impairment will be recruited for this study. Participants' cognitive status will be assessed using the Mini-Mental State Examination (MMSE, <24 cut-off score) and Hopkins Verbal Learning Test (HVLT, <19 cut-off score). Instrumental activities of daily living (IADL) (see below) is used to establish where the cognitive impairment in MCI or dementia. Exclusion criteria will be the following:
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Visual screening | only baseline
  saccade eye movement using eye tracker

SECONDARY OUTCOMES:
Visual Sensitivity test | only baseline
  to measure visual processing speed
driving performance | only baseline
  Hazard perception test (DVLA)
Driving experience survey | only baseline
  driving performance
Corsi Block Span Test | only baseline
  to measure visuospatial working memory
Hopkins Verbal Learning Test | only baseline
  verbal memory
Mini Mental State Examination | only baseline
  Global cognition

CONTACTS AND LOCATIONS:
Locations (1):
- Loughborough University, Loughborough, Leicestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided